CLINICAL TRIAL: NCT01233206
Title: Metformin Addition to Gonadotropins Ovarian Stimulation in High Responder Patients With PCOS Undergoing In-vitro Fertilization
Brief Title: Metformin in High Responder Polycystic Ovary Syndrome (PCOS) Patients Undergoing IVF Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Department of Obstetrics and Gynecology, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04/2010
Record Dates: First submitted 2010-10-08; First posted 2010-11-03 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Infertility; Polycystic Ovary Syndrome (PCOS)
Keywords: PCOS; Polycystic ovary syndrome; Cancelled cycles; OHSS; Infertility
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Patients receiving metformin pretreatment and co-administration
  Interventions: Drug: Metformin
- Control group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo administration

INTERVENTIONS:
Drug: Metformin — Metformin pre-treatment and co-administration
  Arms: Experimental group
Drug: Placebo administration — Placebo pre-treatment and co-administration
  Arms: Control group

SUMMARY:
The use of metformin pre-treatment and co-administration was recently proposed in infertile women affected by polycystic ovary syndrome (PCOS) treated with gonadotropins.

Data from meta-analyses showed that metformin administration significantly reduced the stimulation length and the total dose of gonadotropins used in PCOS women undergoing gonadotropins stimulation for non in-vitro fertilization (IVF) cycles. On the other hand, in IVF cycles metformin was demonstrated to significantly reduce the ovarian hyperstimulation syndrome (OHSS) rate in infertile patients with PCOS treated with gonadotropins.

The metformin regulating effect on the ovarian response was also observed in a randomized controlled trial (RCT) on young non-obese insulin-resistant women with PCOS receiving gonadotropins for mono-ovulation induction. In particular, metformin increased the mono-ovulatory cycles, the duration of stimulation and the amount of gonadotropins used, while it reduced the number of dominant follicles and the estradiol (E2) levels.

The aim of the present study was to evaluate the effect of metformin administration in high responder PCOS patients undergoing gonadotropins ovarian stimulation for IVF cycles.

DETAILED DESCRIPTION:
Infertile young non-obese insulin-resistant patients with PCOS who had a background of the first IVF treatment cycle cancelled because of high risk for OHSS will be enrolled and randomized in two treatment arms.

In their second IVF attempt, the experimental group will receive metformin (500 mg, 3 times daily) pre-treatment for two weeks and co-administration during gonadotropins ovarian stimulation; the control group will be treated with placebo (2 cps daily) pre-treatment and co-administration by using the same schedule of the experimental group. In all patients, ovarian stimulation will be carried out with a personalized step-down gonadotropin in association with a minidose flare-up GnRH agonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* History of one previous cancelled cycle for high-risk of OHSS, or history of moderate/severe OHSS during their previous IVF cycle
* Infertility
* Polycystic ovary syndrome (PCOS)
* insulin resistance
* hyperandrogenism

Exclusion Criteria:

* BMI>30 kg/m2
* age >35 years
* FSH>9UI/L

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Rate of OHSS | one month

SECONDARY OUTCOMES:
Stimulation length | one month
Gonadotropins dose | one month
Dominant follicles on day of ovulation triggering | one month
Ovulation rate | one month
Peak estradiol levels on day of ovulation triggering | one month
Embryo quality | one month
pregnancy rate | one month
multiple pregnancy rate | one month
Live birth rate | ten months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, Principal Investigator — University Magna Graecia; Fulvio Zullo, Study Chair — University Magna Graecia
Locations (1):
- Pugliese" Hospital, Catanzaro, Italy

REFERENCES:
- [Background] Palomba S, Falbo A, Orio F Jr, Manguso F, Russo T, Tolino A, Annamaria C, Dale B, Zullo F. A randomized controlled trial evaluating metformin pre-treatment and co-administration in non-obese insulin-resistant women with polycystic ovary syndrome treated with controlled ovarian stimulation plus timed intercourse or intrauterine insemination. Hum Reprod. 2005 Oct;20(10):2879-86. doi: 10.1093/humrep/dei130. Epub 2005 Jun 15. PMID 15958399
- [Derived] Tso LO, Costello MF, Albuquerque LET, Andriolo RB, Macedo CR. Metformin treatment before and during IVF or ICSI in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD006105. doi: 10.1002/14651858.CD006105.pub4. PMID 33347618
- [Derived] Palomba S, Falbo A, Carrillo L, Villani MT, Orio F, Russo T, Di Cello A, Cappiello F, Capasso S, Tolino A, Colao A, Mastrantonio P, La Sala GB, Zullo F, Cittadini E; METformin in High Responder Italian Group. Metformin reduces risk of ovarian hyperstimulation syndrome in patients with polycystic ovary syndrome during gonadotropin-stimulated in vitro fertilization cycles: a randomized, controlled trial. Fertil Steril. 2011 Dec;96(6):1384-1390.e4. doi: 10.1016/j.fertnstert.2011.09.020. Epub 2011 Oct 7. PMID 21982727